CLINICAL TRIAL: NCT03773133
Title: A Multicentre, Open-Label Phase I/II Study to Evaluate the Safety, Tolerability, Biodistribution and Anti Tumour Activity of 177LU-OPS201 With Companion Imaging 68Ga OPS202 PET/CT in Previously Treated Subjects With Locally Advanced or Metastatic Cancers Expressing Somatostatin Receptor 2 (SSTR2)
Brief Title: Evaluate the Safety, Tolerability, Biodistribution and Anti Tumour Activity of 177LU-OPS201 With Companion Imaging 68Ga-OPS202 PET/CT in Previously Treated Subjects With Locally Advanced or Metastatic Cancers Expressing Somatostatin Receptor 2 (SSTR2)
Acronym: SSTR2+
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: High number of screen failures
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D-FR-01072-002; 2017-005173-39 (EudraCT Number)
Record Dates: First submitted 2018-11-30; First posted 2018-12-12 (Actual); Results first posted 2020-10-30 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Small Cell Lung Cancer and Breast Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Breast Neoplasms | interventions — 177Lu-DOTA-JR11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): i.v. administrations of up to three radioactivity levels of Satoreotide tetraxetan.
  Interventions: Drug: Satoreotide tetraxetan; Drug: Satoreotide trizoxetan

INTERVENTIONS:
Drug: Satoreotide tetraxetan — Radioactivity delivered in 2 administrations (cycles): one loading dose followed by a lower maintenance dose, 6 weeks apart until progression or unacceptable toxicity (up to 4 additional cycles could be administered depending on efficacy and tolerability).
  Other Names: 177Lu-OPS201
Drug: Satoreotide trizoxetan — Imaging companion: 1 administration at screening and one administration at End of core Trial cycle.
  Other Names: 68Ga-OPS202

SUMMARY:
This study consists of two phases. The phase I study is designed to investigate the safety and tolerability of Satoreotide tetraxetan following fractionated i.v. administrations in pre-treated subjects with locally advanced or metastatic cancers expressing sstr2 as identified by Satoreotide trizoxetan Positron Emission Tomography (PET/CT) scans. This phase will encompass both radioactivity escalation and peptide mass dose evaluation. Phase II will assess the efficacy of Satoreotide tetraxetan in subjects in selected indications, in a basket design.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults of Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Histologically confirmed locally advanced or metastatic disease which has progressed during or after, failed to respond to, or for which there is poor tolerability or after a contraindication to available Standard of Care (SoC) treatment options as per the assessment of the investigator; initially, subjects with the disease below may be considered:

  1. Subjects who had Extensive Disease (ED-SCLC) at presentation who have progressed on or after one line standard chemotherapy. If a subject had Limited Disease (LD-SCLC) at presentation and received surgery and/or radiotherapy as first line treatment (with or without chemotherapy) and has localized relapse, further local treatment (such as surgery) should be considered in addition to the chemotherapy options; For subjects with either ED-SCLC or LD-SCLC, if subjects relapse more than 6 months after first-line treatment, re-treatment with their initial regimen is recommended. Subjects may have received prior immunotherapy.
  2. Subjects with Human Epidermal Growth Factor Receptor (HR+)/(HER2-) metastatic BC after a failure of prior SoC-treatments and who have received, if indicated, at least one line of hormonal therapy, Cyclin-dependent kinase (CDK4/6) inhibitor and/or everolimus for advanced or metastatic disease and at least one line of chemotherapy for metastatic disease; subjects with a Breast Cancer (BRCA)-mutated metastatic disease who may have received a Poly adenosine diphosphate ribose polymerase (PARP) inhibitor, if available, are eligible; prior adjuvant hormonal treatment and prior adjuvant chemotherapy are allowed.
* Documented progressive disease (radiological, based on RECIST v1.1) within 3 months prior to first study drug administration. Screening study-related images should be sent to the Imaging core laboratory (ICL).
* Adequate organ function determined within 28 days prior to 177Lu-OPS201 administration, defined as follows:

  * Haematological: white blood cells (WBC) ≥3000/μL, with absolute neutrophil count ≥1000/μL, platelet ≥100,000/μL and haemoglobin ≥9 g/dL (without a need for hematopoietic growth factor or transfusion support).
  * Renal: Estimated glomerular filtration rate (eGFR) ≥55 mL/minute/1.73m2
  * Hepatic: total serum bilirubin ≤2×ULN; aspartate aminotransferase/ alanine aminotransferase ≤2.5×ULN (≤5×ULN if a subject has liver metastases)
* Formalin fixed paraffin embedded tumour sample (archival tumour sample obtained within 1 month prior to concent from the primary or metastatic lesion OR is willing to undergo newly obtained biopsy prior to the first dose of study treatment. Subjects who are unable or do not concent to provide acceptable tissue may not be enrolled unless there has been prior agreement with the sponsor.
* 68Ga OPS202 uptake in the target tissue (a primary tumour, lymph nodes longest diameter on PET/CT as confirmed by a central reader.
* Radiologically, ≥50% matching between the lesions detected on 68Ga OPS202-PET/CT and on 18F-fluorodeoxyglucose (18F-FDG)-PET/CT as confirmed by central reader

Exclusion Criteria:

* Male subjects with BC.
* Unstable central nervous system metastasis
* Centrally located lung tumours that show radiogical evidence (CT or MRI) of either:

  * cavitation or necrosis, or
  * focal invasion for major blood vessels.
* Subjects had received chemotherapy within the previous 4 weeks or had not recovered from adverse events due to chemotherapy. Additional exclusion criteria were previous hemibody external radiotherapy, systemic radiotherapy with radioisotopes within the previous 24 weeks
* Previous chemotherapy within a cycle interval, curative radiotherapy within 4 weeks or palliative radiotherapy within 7 days prior to Investigational radiopharmaceutical product (IRPP) administration.
* Prior treatment with any other investigational medicinal product (IMP) within five half-lives of the previous IMP or within 2 weeks, if the previous compound is a mechanism-based molecularly targeted agent whose half-life is not well characterized and toxicities have not resolved from Grade 2 or higher prior to IRPP administration.
* Any unresolved NCI-CTCAE Grade 2 or higher toxicity (except alopecia and Grade 2 platinum-therapy related neuropathy) from previous antitumour treatment and/or medical/surgical procedures/interventions.
* Nephrectomy, renal transplant or concomitant nephrotoxic therapy putting the subject at high risk of renal toxicity during the study as assessed by the investigator.
* Any significant medical or surgical condition that would affect safety or the assessment of efficacy or the ability of a person to comply with the protocol.
* Any condition that precludes the proper performance of PET and/or SPECT scans, CT scans and/or MRI:

  1. subjects who are not able to tolerate the CT contrast agent.
  2. subjects with metal implants or joint prosthesis (depending on the location, if interferes with the PET and/or CT analysis)
  3. or any other objects that might interfere with the PET and/or CT analysis.
  4. subjects unable to raise arms for prolonged imaging purposes.
  5. subjects unable to lie still for the entire imaging time.
  6. subjects weighing greater than 130 kg (287 lb).
* Pregnant or lactating female. Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 6 months after the last dose of 177Lu-OPS201.
* Male subject who is unwilling to use acceptable method of effective contraception during treatment and through 6 months after the last dose of 177Lu-OPS201.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (8):
- MD Anderson Cancer Center, Houston, Texas, United States
- Medical University of Innsbruck, Innsbruck, Austria
- University Hospital (UZ) Leuven, Leuven, Belgium
- France (2):
  - CHU de Marseille - Hôpital la Timone, Marseille
  - CHU de Bordeaux - Hôpital Haut Lévêque, Pessac
- Universitaetsklinikum Essen, Essen, Germany
- University Hospital Basel, Basel, Switzerland
- Royal Marsden Hospital - Surrey, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase I/II, multicenter, open-label single-arm study of 177Lu-satoreotide tetraxetan therapy with companion diagnostic imaging Gallium-68 (68Ga)-satoreotide trizoxetan (formerly 68Ga-OPS202) positron emission tomography (PET)/computed tomography (CT) was terminated early on 20 November 2019 due to unsuccessful screening.
Pre-assignment Details: Overall, 9 subjects were enrolled of which 8 received the screening investigational imaging product (IIP) 68Ga-satoreotide trizoxetan and 1 did not due to consent withdrawn by subject. None of the subjects received the therapeutic investigational radiopharmaceutical product (IRPP), 177Lu-satoreotide tetraxetan.
Groups:
- Screened Subjects: In the screening period, 8 subjects received a single intravenous (i.v.) injection of IIP, 68Ga-satoreotide trizoxetan with a peptide mass of up to 45 micrograms (ug) and a radioactivity dose range of 150-200 Megabequerel (MBq) for screening purposes. The PET images were acquired at 1-hour post injection and 1 contrast enhanced CT scan was performed.
Period: Overall Study
Arm/Group | Screened Subjects
Started | 8
Received the Screening IIP | 8
Received the Therapeutic IRPP | 0
Completed | 0
Not Completed | 8
Not completed — Screen Failure | 8

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for all subjects who received at least 1 dose of the IIP, 68Ga-satoreotide trizoxetan for screening purposes.
Groups:
- Screened Subjects: In the screening period, 8 subjects received a single i.v. injection of IIP, 68Ga-satoreotide trizoxetan with a peptide mass of up to 45 ug and a radioactivity dose range of 150-200 MBq for screening purposes. The PET images were acquired at 1-hour post injection and 1 contrast enhanced CT scan was performed.
Arm/Group | Screened Subjects
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Cumulative Activity - Phase I
Time Frame: From Day 1 (first administration of 177Lu-satoreotide tetraxetan) up to 6 weeks after the second administration; no longer applicable due to early study termination.
Population: No efficacy data was collected since none of the subjects received the IRPP, 177Lu-satoreotide tetraxetan.
Groups:
- All Subjects - Phase I: In the core treatment period of Phase I, eligible subjects were to receive up to 2 i.v. administrations of 177Lu-satoreotide tetraxetan. A range of cumulative radioactivities from 9 to 12.9 Gigabecquerels of 177Lu-satoreotide tetraxetan, fractionated into 2 administrations 6 weeks apart, were planned to be tested.
Arm/Group | All Subjects - Phase I
Number analyzed (Participants) | 0

2. Primary Outcome: Objective Response Rate Over the Two Treatment Cycles - Phase II
Time Frame: 6 weeks after each administration of 177Lu-satoreotide tetraxetan during the core study or at occurrence of first clinical signs of disease progression as determined by the investigator, up to 90 days; no longer applicable due to early study termination.
Population: No efficacy data was collected since none of the subjects received the IRPP, 177Lu-satoreotide tetraxetan.
Groups:
- All Subjects - Phase II: Subjects were to receive the recommended Phase II 177Lu-satoreotide tetraxetan treatment regimen based on the dose-response and exposure-response analyses of Phase I. It was expected that 2 treatment cycles of 177Lu-satoreotide tetraxetan would be administered in subjects enrolled in Phase II.
Arm/Group | All Subjects - Phase II
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were assessed after first administration of the IIP, 68Ga-satoreotide trizoxetan, until the data cut-off for study termination (maximum of 21 weeks).
Groups:
- 68Ga-satoreotide Trizoxetan Safety Population: The 68Ga-satoreotide trizoxetan safety population included all subjects who received at least 1 dose of 68Ga-satoreotide trizoxetan.
Arm/Group | 68Ga-satoreotide Trizoxetan Safety Population
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 68Ga-satoreotide Trizoxetan Safety Population (N=8)
Iodine allergy (Immune system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to unsuccessful screening and not due to subjects' safety. No outcomes measures were evaluated as no subjects received the therapeutic IRPP, 177Lu-satoreotide tetraxetan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT03773133/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT03773133/SAP_001.pdf